CLINICAL TRIAL: NCT03180996
Title: A Prospective, Global, Multicentre, Real World Outcome Study of Fenestrated Endovascular Aneurysm Repair Using the Fenestrated Anaconda™ Device
Brief Title: Global Fenestrated Anaconda Clinical STudy
Acronym: Global FACT
Status: Active, not recruiting | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: FACT-001
Record Dates: First submitted 2017-05-24; First posted 2017-06-08 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: FEVAR; Fenestrated; Endovascular; AAA; Custom device
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Vascutek Fenestrated Anaconda™ Custom AAA Stent Graft System — Fenestrated Endovascular Aortic Repair (FEVAR)

SUMMARY:
This study is a prospective non-interventional, multi-centre study of the Vascutek Fenestrated Anaconda™ system, and is essentially a post-market study. The Vascutek Fenestrated Anaconda™ system is a custom made device used for the treatment of Abdominal Aortic Aneurysm.

DETAILED DESCRIPTION:
Abdominal Aortic Aneurysm (AAA) is a life threatening disease. Endovascular repair of infrarenal abdominal aortic aneurysms (EVAR) has replaced open surgical repair as the standard of care treatment for most patients. Endovascular repair offers several benefits over open surgical repair, including: less invasive procedure, faster recovery, lower morbidity and lower early post-operative mortality. The configuration of vascular anatomy is important to the successful placement and subsequent performance of infrarenal EVAR devices. In particular aortic neck angulation and length are important for the success of EVAR. Challenging necks with an aortic diameter ≥28 mm, angulation ≥60°, length <10mm, circumferential thrombus, reversed tapered configuration or neck with bulging, make it more difficult to oppose the endograft to the aortic wall and are related to an increased risk of type Ia endoleak and reinterventions. In order to overcome these issues, fenestrated and branched stent grafts have been developed. Fenestrated and branched endovascular aneurysm repair is now a routinely utilised procedure in the treatment of complex aortic aneurysm anatomy, especially in patients unsuitable for open surgical repair.

The Fenestrated Anaconda™ device (Vascutek Ltd, Glasgow, Scotland, UK) has been commercially available since 2010. The Fenestrated Anaconda™ device has potential advantages over other FEVAR devices, since it can be repositioned after deployment, has a magnet-assisted limb cannulation, and the device contains less metal, allowing a better view of the radiological markers on the device during intra-operative imaging. Additionally, the potential to position fenestrations anywhere in the main body is unrestricted due to the absence of other stent structures.

This prospective, real world study of the Fenestrated Anaconda™ device will provide insight into both the short and long term clinical outcomes of the device. An attempt will be made to identify predictors of success or failure, and this study will help to identify patients that are likely to benefit from repair and improve results. The effect of FEVAR on post-operative patient reported quality of life will be assessed. In addition, the study will provide insight into the potential decline in renal function after FEVAR, a well-known concern after both EVAR and FEVAR.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the criteria below in order to be eligible for inclusion in the study -

1. Patient is aged 18 years or over on the date of consent
2. Patient is willing and able to comply with all study procedures and study follow-up visits
3. Patient is willing and able to give written informed consent to participate in study
4. Patient has a juxtrarenal or suprarenal abdominal aortic aneurysm (AAA) with maximum sac diameter ≥ 5.5cm, or an AAA ≥ 4.5 cm which has increased by > 1.0 cm in the past year
5. Patient is anatomically suitable for a bifurcated Fenestrated Anaconda™ device

NOTE: Both the treating Investigator and the Manufacturer must agree that the proposed patient's anatomy is suitable for treatment using the Fenestrated Anaconda™ device. Where the Investigator proposes that the patient anatomy is suitable and the Manufacturer subsequently disagrees, the patient will be recorded as a screen failure and deemed not eligible for the study.

Exclusion Criteria:

Any patient who meets any of the criteria below will be excluded from participation in the study -

1. Patient has a life expectancy < 2 years, as judged by the Investigator
2. Patient has psychiatric or other condition that in the opinion of the Investigator may limit their ability to comply with study procedures
3. Patient is participating in another clinical study which in the opinion of the Investigator could influence the outcomes of this study
4. Patient has a known allergy to any device component (polyester, nitinol, nickel)
5. Patient has a coagulopathy or uncontrolled bleeding disorder
6. Patient has a ruptured, leaking or mycotic aneurysm
7. Patient has a serum creatinine (S-Cr) level > 2.0 mg/dL (177 µmol/L)
8. Patient has had CVA or MI within three months of enrolment or treatment
9. Patient has a connective tissue disease (e.g. Marfan Syndrome)
10. Patient has had a previously inserted endovascular stent in the abdominal aorta
11. Patient is pregnant (female of childbearing potential only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a juxtrarenal or suprarenal abdominal aortic aneurysm, including those aneurysms with very short neck or no neck, who require endovascular repair of their aneurysm and whose aneurysm is suitable for treatment using a custom made Vascutek Fenestrated Anaconda™ device will be recruited. This is a non-interventional study and therefore only patients who would normally receive this device as part of standard treatment at the participating institute will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who experience Treatment Success. | 1 year post-procedure
  Treatment success is defined as freedom from the following: Type I and III endoleak; stent graft migration; AAA enlargement; AAA rupture; conversion to open surgery; non-patent endoluminal grafts and/or significant twists, kinks or obstruction; aneurysm-related patient death.

CONTACTS AND LOCATIONS:
Overall Officials: Clark J Zeebregts, MD, PhD, Prof, Principal Investigator — Universitair Medisch Centrum Groningen (UMCG), Netherlands; Michel MPJ Reijnen, MD, PhD, Prof, Principal Investigator — Rijnstate Hospital, Arnhem, Netherlands
Locations (11):
- Australia (2):
  - Epworth Richmond Private Hospital, Melbourne, Victoria
  - Hollywood Medical Centre, Perth, Western Australia
- Wilhelminenspital, Vienna, Austria
- Peter Lougheed Centre, Calgary, Alberta, Canada
- Netherlands (4):
  - Rijnstate Hospital, Arnhem
  - Medisch Spectrum Twente (MST), Enschede
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Antonius Ziekenhuis, Nieuwegein
- United Kingdom (3):
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Frimley Park Hospital, Camberley
  - Imperial College, St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No